CLINICAL TRIAL: NCT07080801
Title: Study on the Safety and Efficacy of RAG-21 in the Treatment of Amyotrophic Lateral Sclerosis Patients With FUS Gene Mutations
Acronym: RAG-21-FUS-ALS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice-President of Beijing Tiantan Hospital,Chief Scientist of Neurology Center, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-A-2025021
Record Dates: First submitted 2025-07-06; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: RAG-21; FUS gene mutations
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAG-21 (Experimental)
  Interventions: Drug: RAG-21

INTERVENTIONS:
Drug: RAG-21 — Intrathecal bolus administration of RAG-21 will be initiated at a dose of 120 mg, prepared with a dedicated solvent into a 10 mL sterile aqueous solution. Dosing will occur every 2 weeks, with the dose escalating to 180 mg after 3 administrations. Subsequently, the dosing interval will be extended to every 4 weeks. The investigator will then select an optimal dose from the completed dose cohorts or continue dose escalation until the maximum tolerated dose (MTD) is reached, with a predefined maximum dose of 210 mg. For continued treatment, the investigator-determined optimal dose will be administered as a fixed dose every 4 weeks, with a total treatment duration of 6 months (8 administrations).

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a chronic progressive neurodegenerative disease that remains incurable, with limited existing therapies or drugs available. Familial ALS can be caused by mutations in various genes. In Asia, mutations in the FUS gene are relatively common among early-onset familial ALS patients. Reducing the levels of toxic FUS protein may be an effective therapeutic approach for such ALS patients without causing side effects.

RAG-21 is a small interfering ribonucleic acid (siRNA) with a molecular weight of 20 kDa. Through the RNA interference mechanism, it targets the FUS gene, recognizes the corresponding mRNA, and mediates its degradation, thereby downregulating FUS gene expression and reducing toxic FUS protein levels. Accordingly, this project plans to conduct a single-center, dose-escalation clinical study aimed at evaluating the safety, tolerability, and pharmacokinetics of intrathecal bolus administration of RAG-21 in ALS patients carrying FUS gene mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, gender unlimited.
2. Clearly identify amyotrophic lateral sclerosis (ALS) patients with FUS gene mutations (known FUS mutation sites and reported disease progression).
3. Forced vital capacity (FVC) during screening period ≥ 50% of expected lung capacity.
4. ALS patients diagnosed according to the Gold Coast criteria (2020) with limb-onset weakness.
5. The patient or their legal representative clearly understands and voluntarily participates in the study and signs an informed consent form.
6. The subjects (including male subjects) have no family planning throughout the entire study and within 3 months after, voluntarily take effective contraceptive measures and without any plans to donate sperm or ovum.

Exclusion Criteria:

1. FUS mutation sites located within nucleotides 928-970 (calculated from the translation of FUS protein).
2. Patients who have previously received or are currently receiving Ulefnersen treatment.
3. Human immunodeficiency virus (HIV) test positive or positive test history.
4. Patients with active hepatitis C or hepatitis B infection.
5. Other experimental drugs used within one month or within five drug half-lives.
6. Lumbar diseases and deformities.
7. ALS with bulbar-onset symptoms, or suffering from other diseases known to be related to motor neuron dysfunction, which may confuse or blur the diagnosis of ALS.
8. Other psychiatric disorders diagnosed according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnostic criteria, or obvious suicidal intentions.
9. Combined with severe liver dysfunction, renal dysfunction, or severe heart dysfunction (severe liver dysfunction refers to alanine aminotransferase (ALT) value ≥ 2.0 times the upper limit of normal value or aspartate aminotransferase (AST) value ≥ 2.0 times the upper limit of normal value; severe renal dysfunction refers to creatinine (CRE) ≥ 1.5 times the upper limit of normal value or estimated glomerular filtration rate (eGFR) < 40mL/min/1.73m^2; severe heart dysfunction refers to New York College of Cardiology (NYHA) 3-4 levels).
10. Permanent and sustained dependence on ventilator assisted ventilation.
11. History of combined alcohol and drug abuse.
12. Pregnant, lactating, or potentially pregnant patients, as well as those planning to conceive.
13. Patients participating in other clinical trials or applying other biologics, drugs, or devices under study.
14. Patients who have received any vaccination within 28 days.
15. Those who can't complete follow-up due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
AE&SAE | 15±1, 29±2, 57±3, 85±3, 113±3, 141±3, 169±3, 197±7days after treatment
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) after RAG-21 treatment.

IPD SHARING:
Plan to Share IPD: No